CLINICAL TRIAL: NCT02350153
Title: National Swedish Study in Cushing´s Disease Incidence and Outcomes
Brief Title: Cushing´s Disease Epidemiology in Sweden
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: NSSCDIO
Record Dates: First submitted 2014-12-05; First posted 2015-01-29 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Cushing Disease
Keywords: Mortality; Morbidity; Incidence; Prevalence
MeSH Terms: conditions — Pituitary ACTH Hypersecretion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with verified Cushing's Disease: Patients with verified Cushing's Disease

SUMMARY:
The purpose of this study is to study since 1987 all patients diagnosed with CD in Sweden and determine their outcomes including mortality. A secondary objective is to focus on patients in remission and identify determinants of their different outcomes.

DETAILED DESCRIPTION:
This study is a retrospective nationwide study of all patients in Sweden with diagnosis CD between 1987 and 2013 were baseline data at diagnosis, information about the different treatments and follow-up data is going to be obtained by reviewing patients' medical journals. This information as well as the exact diagnose criteria for each patient are going to be extracted by Endocrinologists in all University Hospitals in Sweden. An expert group at the Sahlgrenska University Hospital in Gothenburg will put together the data.By the use of the Swedish Personal Number, the investigators are going to obtain information about both patients' and background population co-morbidities which have been collected in the different Swedish Registers.

Primary aim:

To study mortality of CD in Sweden.

Secondary aims:

1. To study the influence of CD on myocardial infarction
2. To study the influence of CD on stroke
3. To study the influence of CD on cancer
4. To study the influence of CD on hip fracture risk
5. To study incidence and prevalence of CD in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* All patients registered with Cushing's Disease in Sweden since 1987 in the statistical database for in- and out-patients, at the Swedish National Board of Health and Welfare will be included in the study.

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with confirmed CD diagnosis in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2013-09; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Mortality | From date of diagnosis until the last day of December 2014 or date of death from any cause, whichever came first, assessed up to 20 years.
  If event (death) has been occured during the observation period. Data obtained by the Swedish Cause Of Death Register (Swedish Board of Health and Welfare)

SECONDARY OUTCOMES:
influence of Cushing's Disease on myocardial infarction | From date of diagnosis until the last day of December 2014 or date of death from any cause, whichever came first, assessed up to 20 years
  If event (myocardial infarction) has been occured during the observation period.Data obtained by the Swedish Register of In- and Out-patient Diagnoses (Swedish Board of Health and Welfare)
influence of Cushing's Disease on stroke | From date of diagnosis until the last day of December 2014 or date of death from any cause, whichever came first, assessed up to 20 years
  If event (stroke) has been occured during the observation period.Data obtained by the Swedish Register of In- and Out-patient Diagnoses (Swedish Board of Health and Welfare)
influence of Cushing's Disease on cancer | From date of diagnosis until the last day of December 2014 or date of death from any cause, whichever came first, assessed up to 20 years
  If event (cancer) has been occured during the observation period.Data obtained by the Swedish Register of Cancer Diagnoses (Swedish Board of Health and Welfare)
influence of Cushing's Disease on hip fracture risk | From date of diagnosis until the last day of December 2014 or date of death from any cause, whichever came first, assessed up to 20 years
  If event (hip fracture) has been occured during the observation period.Data obtained by the Swedish Register of Hip Fractures (Swedish Board of Health and Welfare)
incidence of Cushing's Disease in Sweden | Assessed up to 20 years.
  Validation of Data obtained by The Swedish Board of Health and Welfare by reviewing all patients' journals
prevalence of Cushing's Disease in Sweden | Assessed up to 20 years.
  Validation of Data obtained by The Swedish Board of Health and Welfare by reviewing all patients' journals

CONTACTS AND LOCATIONS:
Overall Officials: Gudmundur Johannsson, Professor, Principal Investigator — Vastra Gotaland Region, Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided